CLINICAL TRIAL: NCT03448952
Title: Incidence and Risk Factors for Neonatal Thrombocytopenia Among Newborns Admitted to Neonatal Intensive Care Unit of Assiut University Children Hospital
Brief Title: Neonatal Thrombocytopenia Among Newborns Admitted to Neonatal Intensive Care Unit
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sylvia Elzek (Other)
Responsible Party: Sponsor-Investigator, Sylvia Elzek, principle investigator, Assiut University
Organization: Assiut University (Other)
Other Study IDs: IRNT
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Thrombocytopenia Neonatal
MeSH Terms: conditions — Thrombocytopenia, Neonatal Alloimmune

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Thrombocytopenia is diagnosed when platelet count is lower than 150,000 U/L, it is a common hemostatic problem in neonatal intensive care units According to platelets count, it is classified into mild thrombocytopenia with platelet count 100,000 to 150,000 U/L, moderate thrombocytopenia with platelet count 50,000 to 100,000 U/L and severe thrombocytopenia that have platelet count less than or equal to 50,000 U/L.

DETAILED DESCRIPTION:
Platelets are seen under microscope as small anucleated fragments of megakaryocytes that circulate in the blood as discs with an average volume of about 7.5 fimtolitre , 14 times smaller than erythrocytes. Platelets count in premature infant is slightly lower than that of healthy term infant but is still within the normal range (150,000 to 450,000 unit/ litre ).

The most common risk factors for thrombocytopenia are

1. Sepsis: Thrombocytopenia is a frequent problem in neonatal sepsis and is among the most predictive, independent risk factors for sepsis-associated mortality
2. Low birth weight: It is recorded that thrombocytopenia was more common among the smallest patients; 85% incidence among those ⩽800 gram, 60% among those 801 to 900 gram, and 53% among those 901 to 1000 gram
3. Perinatal asphyxia: Thrombocytopenia occurred in 31% of neonates with asphyxia versus 5% of matched non asphyxiated controls admitted to a neonatal intensive care unit
4. Prematurity: In a normal pregnancy, the fetal platelet count reaches adult levels (150-450 × 106/ millilitre) by the second trimester of pregnancy. Thrombocytopenia , defined as less than 150,000/ millilitre, occurs in 18 to 40% of all preterm neonates (gestational age <37 weeks) admitted to neonatal intensive care units

ELIGIBILITY:
Inclusion Criteria:

1. newborn (term and preterm, inborn or out born) aged from 1-28 day
2. platelet count below one hundred and fifty thousands unit/liter

Exclusion Criteria:

1. Infant above 28 days old.
2. Newborns have platelet count one hundred and fifty thousands unit/liter

Exclusion Criteria:

Ages: 1 Hour to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study will include all newborns with thrombocytopenia either preterm or full term, inborn or out born cases who admitted to neonatal intensive care unit of Assiut University Children Hospital through one year.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
incidence of thrombocytopenia in newborn admitted to neonatal intensive care unit of Assiut University Children Hospital. | 1-28 day after birth
  measure the incidence of thrombocytopenia in newborn admitted to neonatal intensive care unit of Assiut University Children Hospital.
risk factors of of thrombocytopenia in newborn admitted to neonatal intensive care unit of Assiut University Children Hospital. | 1-28 day after birth
  detect the risk factors of thrombocytopenia in newborn admitted to neonatal intensive care unit of Assuit University Children Hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Safwat Abd ElAziz, MD, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided